CLINICAL TRIAL: NCT01863472
Title: Catheter Ablation of Drug-refractory Persistent Atrial Fibrillation With the HeartLight(TM) Laser Balloon in Comparison With Irrigated Radiofrequency Current Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boris Schmidt (Other)
Responsible Party: Sponsor-Investigator, Boris Schmidt, Arzt für Kardiologie, Cardioangiologisches Centrum Bethanien
Organization: Cardioangiologisches Centrum Bethanien (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF20/13 Version 03
Record Dates: First submitted 2013-05-19; First posted 2013-05-29 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HeartLight(TM) Laser Balloon (Active Comparator): Safety and efficacy of pulmonary vein isolation using the HeartLight(TM) Laser Balloon (endoscopically guided ablation)
  Interventions: Device: HeartLight(TM) Laser Balloon
- irrigated radiofrequency current ablation (Active Comparator): Safety and efficacy of pulmonary vein isolation using the irrigated radiofrequency current ablation
  Interventions: Device: irrigated radiofrequency current ablation

INTERVENTIONS:
Device: HeartLight(TM) Laser Balloon — With the HeartLight(TM) Laser Balloon pulmonary vein isolation is done endoscopically guided
  Arms: HeartLight(TM) Laser Balloon
Device: irrigated radiofrequency current ablation — The irrigated radiofrequency current ablation is used for pulmonary vein isolation
  Arms: irrigated radiofrequency current ablation

SUMMARY:
Aim of the study is to compare the safety and efficacy of pulmonary vein isolation using the endoscopic ablation system in comparison to irrigated radiofrequency current ablation in patients with drug-refractory persistent atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years
* persistent atrial fibrillation
* failure of at least one antiarrhythmic drug
* others

Exclusion Criteria:

* contraindications for pulmonary vein isolation (PVI)
* previous PVI attempts
* inability to be treated with oral anticoagulation
* presence of intracardiac thrombi
* pregnancy
* others

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-06; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Documented recurrence of atrial fibrillation or any atrial tachyarrhythmia >30 seconds | between day 90 and 365 days after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Boris Schmidt, Dr., Principal Investigator — Cardioangiologisches Centrum Bethanien
Locations (6):
- Na Homolce Hospital, Prague, Czechia
- Germany (4):
  - Herz- und Gefäß-Klinik GmbH Bad Neustadt, Bad Neustadt an der Saale, Bavaria
  - Rheinische Friedrich-Wilhelms-Universität Bonn, Bonn, North Rhine-Westphalia
  - Cardioangiologisches Centrum Bethanien, Frankfurt am Main
  - Städtisches Klinikum Karlsruhe, Medizinische Klinik IV, Karlsruhe
- Hospital Universitari i Politecnic La Fe, Valencia, Spain

REFERENCES:
- [Derived] Schmidt B, Neuzil P, Luik A, Osca Asensi J, Schrickel JW, Deneke T, Bordignon S, Petru J, Merkel M, Sediva L, Klostermann A, Perrotta L, Cano O, Chun KRJ. Laser Balloon or Wide-Area Circumferential Irrigated Radiofrequency Ablation for Persistent Atrial Fibrillation: A Multicenter Prospective Randomized Study. Circ Arrhythm Electrophysiol. 2017 Dec;10(12):e005767. doi: 10.1161/CIRCEP.117.005767. PMID 29217521